CLINICAL TRIAL: NCT05464550
Title: Role of Self-focused Attention in Depression
Acronym: RFASD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Henri Laborit (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2021-A01098-33
Record Dates: First submitted 2022-04-21; First posted 2022-07-19 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Eye tracking (Experimental): Utilisation of a eye tracker on a screen.
  Interventions: Behavioral: Eye tracker

INTERVENTIONS:
Behavioral: Eye tracker — Eye movements on a screen are captured with an eye tracker during a repeated measures before/after a directed autobiographical recall.

SUMMARY:
Using a task measuring the tracking of eye movements, the aim of this study is to demonstrate that individuals suffering from depression focus their attention more on their reflection in the screen after recalling a failure (and this all the more so as their depressive symptomatology is strong) .

ELIGIBILITY:
Inclusion Criteria:

* patients with depressive disorders according to the Diagnostic and statistical Manual of Mental Disorders (DSM-V) criteria
* Men or women, aged 18 to 60
* patients without mental impairment
* patients without neurological impairment (epilepsy, encephalopathy, head trauma)
* patients with a sufficient command of French
* free patients, without guardianship or curators or subordination
* patients benefiting from coverage by a social security scheme or benefiting from it through a third party in accordance with the French law on biomedical research
* obtaining oral non-objection by the patient after clear and honest information about the study
* Patient with normal or corrected vision without rigid contact lenses

Exclusion Criteria:

* patients with an intelligence quotient < 70
* patients aged < 18 years or > 60 years
* patients with mental impairment
* patients with neurological impairment (epilepsy, encephalopathy, head trauma)
* patients who do not speak French well enough
* patients hospitalized under duress
* patients without social security
* Patient wearing rigid contact lenses

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-12-08 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-06-16 (Actual)

PRIMARY OUTCOMES:
Percentage of time | through study completion, an average of 10 months.
  Average percentage of time spent on the area of a reflective black computer screen after and before remembering a failure. The area of interest encompasses the reflection of the patient's face, without his attention being explicitly drawn to this area.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Henri Laborit, Poitiers, France

IPD SHARING:
Plan to Share IPD: No